CLINICAL TRIAL: NCT05003453
Title: The Effectiveness of a Topical Palmitoylethanolamide Formulation (Levagen+) for Reducing the Symptoms of Eczema Versus a Comparator
Brief Title: The Effectiveness of a Topical Palmitoylethanolamide (PEA) Formulation (Levagen+) for Reducing Symptoms of Eczema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEA-XMA-20
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-08

CONDITIONS: Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — palmidrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.5% Palmitoylethanolamide (PEA) sold as Levagen+ (Experimental): Investigational product will be provided as a topical cream containing 1.5% PEA and participants will be asked to apply to their affected site 2 times daily for 4 weeks. Cream should be applied liberally (as you would a moisturiser cream) such to coat the affected area and absorb into the skin.
  Interventions: Drug: 1.5% Palmitoylethanolamide (PEA) sold as Levagen+
- Placebo comparator (Placebo Comparator): A comparator placebo moisturiser cream (an unscented moisturizing base cream) will be provided and applied in the same manner as the active ingredient group. Participants will be asked to apply to their affected site 2 times daily for 4 weeks. Cream should be applied liberally (as you would a moisturiser cream) such to coat the affected area and absorb into the skin.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: 1.5% Palmitoylethanolamide (PEA) sold as Levagen+ — A topical cream containing 1.5% PEA applied to the affected site 2-times daily, liberally to coat and cover affected area.
  Other Names: PEA, Levagen+
  Arms: 1.5% Palmitoylethanolamide (PEA) sold as Levagen+
Drug: Placebo Comparator — A comparator placebo topical moisturiser cream (an unscented moisturising base cream) applied to the affected site 2 times daily, liberally to coat and cover affected area.
  Other Names: Moisturising cream
  Arms: Placebo comparator

SUMMARY:
This is a double blind, randomised, non-clinical study with 2 groups (1 investigational group and 1 comparator group) aiming to assess the effectiveness of PEA for reducing eczema severity compared to a base comparator moisturiser in healthy adults aged over 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18)
* Suffering from atopic eczema with symptoms of redness, dry skin, scaling and/or itchiness on hands or arms
* Otherwise healthy
* Able to provide informed consent

Exclusion Criteria:

* Active allergic skin responses
* Unstable or serious illness (eg kidney, liver, GIT, heart conditions, diabetes, mood disorders, cancer)
* Use of immunosuppressive medication within the last 3 months
* Pregnant or lactating women
* Smokers
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in active or comparator formula

  * An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Eczema area and severity index (SA-EASI) | Baseline prior to commencement, Week 2 and Week 4
  Change in eczema area and severity index (SA-EASI)

SECONDARY OUTCOMES:
Change in itchiness (pruritus numerical rating scale) | Baseline prior to commencement, Week 2 and Week 4
  Change in self-reported itchiness (pruritus numerical rating scale). Minimum value = 0, no pruritus. Maximum value = 10, Very severe pruritus.
Change in topical anti-inflammatory use | Baseline prior to commencement, Week 2 and Week 4
  Change in self-reported topical anti-inflammatory use
Patient eczema self assessment (Patient Orientated Eczema Measure) | Baseline prior to commencement, Week 2 and Week 4
  Improvement in POEM. Minimum value 0 - clear or almost clear, Maximum value 28 - Very severe eczema
Change in Quality of Life (DQOL) | Baseline prior to commencement, Week 2 and Week 4
  Change in quality of life questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: David Briskey, PhD, Principal Investigator — The University of Queensland
Locations (1):
- RDC Global Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Rao A, Moussa AA, Erickson J, Briskey D. Efficacy of Topical Palmitoylethanolamide (Levagen+) for the Management of Eczema Symptoms: A Double-Blind, Comparator-Controlled, Randomized Clinical Trial. Skin Pharmacol Physiol. 2023;36(6):288-295. doi: 10.1159/000536670. Epub 2024 Feb 26. PMID 38408443